CLINICAL TRIAL: NCT03383042
Title: A Randomized, Open-label, Placebo- and Active- Controlled, Single and Multiple Ascending Dose Phase I Clinical Trial to Investigate the Safety, Tolerability and Pharmacokinetics and Pharmacodynamics of JP-1366 Oral Administration in Healthy Male Subjects
Brief Title: Clinical Trial to Investigate the Safety, Tolerability and Pharmacokinetics and Pharmacodynamics of JP-1366 Oral Administration in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jeil Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JP-1366-101-FIH
Record Dates: First submitted 2017-12-18; First posted 2017-12-26 (Actual); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Anti-Ulcer Agents
MeSH Terms: interventions — mycophenolic adenine dinucleotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Cohort 1 (Experimental): Single-ascending cohort 1
  Interventions: Drug: Cohort 1 (JP-1366 A mg)
- Cohort 2 (Experimental): Single-ascending cohort 2
  Interventions: Drug: Cohort 2 (JP-1366 B mg)
- Cohort 3 (Experimental): Single-ascending cohort 3
  Interventions: Drug: Cohort 3 (JP-1366 C mg)
- Cohort 4 (Experimental): Single-ascending cohort 4
  Interventions: Drug: Cohort 4 (JP-1366 D mg)
- Cohort 5 (Experimental): Single-ascending cohort 5
  Interventions: Drug: Cohort 5 (JP-1366 E mg)
- Cohort 6 (Experimental): Multiple-ascending cohort 1
  Interventions: Drug: Cohort 6 (JP-1366 F mg)
- Cohort 7 (Experimental): Multiple-ascending cohort 2
  Interventions: Drug: Cohort 7 (JP-1366 G mg)
- Cohort 8 (Experimental): Multiple-ascending cohort 3
  Interventions: Drug: Cohort 8 (JP-1366 H mg)
- Cohort 9 (Experimental): Multiple-ascending cohort 4
  Interventions: Drug: Cohort 9 (JP-1366 I mg)

INTERVENTIONS:
Drug: Cohort 1 (JP-1366 A mg) — Drug: JP-1366 A mg or JP-1366 Placebo or Esomeprazole 40 mg
  Other Names: SAD
  Arms: Cohort 1
Drug: Cohort 2 (JP-1366 B mg) — Drug: JP-1366 B mg or JP-1366 Placebo or Esomeprazole 40 mg
  Other Names: SAD
  Arms: Cohort 2
Drug: Cohort 3 (JP-1366 C mg) — Drug: JP-1366 C mg or JP-1366 Placebo or Esomeprazole 40 mg
  Other Names: SAD
  Arms: Cohort 3
Drug: Cohort 4 (JP-1366 D mg) — Drug: JP-1366 D mg or JP-1366 Placebo or Esomeprazole 40 mg
  Other Names: SAD
  Arms: Cohort 4
Drug: Cohort 5 (JP-1366 E mg) — Drug: JP-1366 E mg or JP-1366 Placebo or Esomeprazole 40 mg
  Other Names: SAD
  Arms: Cohort 5
Drug: Cohort 6 (JP-1366 F mg) — Drug: JP-1366 F mg or JP-1366 Placebo or Esomeprazole 40 mg
  Other Names: MAD
  Arms: Cohort 6
Drug: Cohort 7 (JP-1366 G mg) — Drug: JP-1366 G mg or JP-1366 Placebo or Esomeprazole 40 mg
  Other Names: MAD
  Arms: Cohort 7
Drug: Cohort 8 (JP-1366 H mg) — Drug: JP-1366 H mg or JP-1366 Placebo or Esomeprazole 40 mg
  Other Names: MAD
  Arms: Cohort 8
Drug: Cohort 9 (JP-1366 I mg) — Drug: JP-1366 I mg or JP-1366 Placebo or Esomeprazole 40 mg
  Other Names: MAD
  Arms: Cohort 9

SUMMARY:
Clinical trial to investigate the safety, tolerability and pharmacokinetics and pharmacodynamics of JP-1366 oral administration in healthy male subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males aged between 19 and 50 at screening
* Weight is between 55 and 90 kg and BMI is between 18.0 and 27.0
* Those who are adequate to be subjects in this study upon judgment of the investigator after physical examination, clinical laboratory test, examination by interview, etc

Exclusion Criteria:

* Subject has clinical significant liver, kidney, nervous system, respiratory, endocrine, hematology and oncology, cardiovascular, urinary, and mental diseases or past history
* Subject has gastrointestinal diseases or past history of gastrointestinal diseases (gastrointestinal ulcer, gastritis, gastrospasm, gastroesophageal reflux, Crohn's disease etc.) that may affect safety and pharmacokinetic/pharmacodynamic evaluation of study drug, and those who have past history of gastrointestinal surgery (however, except simple appendectomy and herniotomy)
* Subject has been Helicobacter pylori positive
* AST (SGOT) and ALT (SGPT) > 1.5 times to the upper limit of the normal range in screening including additional examinations prior to randomization
* Subject has anatomical disability in insertion and maintenance of pH meter catheter

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 115 (Actual)
Dates: Start 2017-12-22 (Actual); Primary Completion 2018-11-23 (Actual); Study Completion 2019-04-05 (Actual)

PRIMARY OUTCOMES:
Cmax | Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24 and 48 hours post-dose
  SAD endpoint
AUClast | Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24 and 48 hours post-dose
  SAD endpoint
AUCinf | Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24 and 48 hours post-dose
  SAD endpoint
tmax | Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24 and 48 hours post-dose
  SAD endpoint
t1/2 | Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24 and 48 hours post-dose
  SAD endpoint
Cmax,ss | Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24h post-dose, Day 3-6, pre-dose, Day 7 pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24 and 48 hour post-dose
  MAD endpoint
Cmin,ss | Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24h post-dose, Day 3-6, pre-dose, Day 7 pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24 and 48 hour post-dose
  MAD endpoint
Cav,ss | Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24h post-dose, Day 3-6, pre-dose, Day 7 pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24 and 48 hour post-dose
  MAD endpoint
AUCτ | Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24h post-dose, Day 3-6, pre-dose, Day 7 pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24 and 48 hour post-dose
  MAD endpoint
tmax,ss | Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24h post-dose, Day 3-6, pre-dose, Day 7 pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24 and 48 hour post-dose
  MAD endpoint
t1/2 | Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24h post-dose, Day 3-6, pre-dose, Day 7 pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24 and 48 hour post-dose
  MAD endpoint
Percentage of total time that the intragastric pH was above 4 | 0-24 hours(Day -1), 0-24 hours(Day 1)
  SAD
Percentage of total time that the intragastric pH was above 4 | 0-24 hours (Day -1), 0-24 hours (Day 1), 0-24 hours (Day 7)
  MAD
Serum gastrin concentration | Pre-dose, 2, 4, 6, 8, 12h post-dose, Day 1 pre-dose, 2, 4, 6, 8, 12, 24, 48h post-dose
  SAD
Serum gastrin concentration | Pre-dose, 2, 4, 6, 8, 12h post-dose, Day 1 pre-dose, 2, 4, 6, 8, 12, 24h post-dose, Day 4 pre-dose, Day 6 pre-dose, Day 7 pre-dose, 2, 4, 6, 8, 12, 24, 48h post-dose
  MAD

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital(SNUH), Seoul, Jongno-Gu, South Korea

IPD SHARING:
Plan to Share IPD: No